CLINICAL TRIAL: NCT04173637
Title: A Randomized, Double-blinded, Placebo-controlled, Phase IIb Clinical Study of AK101 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Clinical Study of AK101 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK101-301
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Plaque Psoriasis
Keywords: IL12/23

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AK101 45mg every 8 weeks (Experimental): AK101 45mg on Week 0 and 4 administered subcutaneously followed by AK101 45mg administered subcutaneously every 8 weeks
  Interventions: Biological: AK101
- AK101 45mg - every 12 weeks (Experimental): AK101 45mg on Week 0 and 4 administered subcutaneously followed by AK101 45mg administered subcutaneously every 12 weeks
  Interventions: Biological: AK101
- AK101 90mg - every 8 weeks (Experimental): AK101 90mg on Week 0 and 4 administered subcutaneously followed by AK101 90mg administered subcutaneously every 8 weeks
  Interventions: Biological: AK101
- AK101 90mg -every 12 weeks (Experimental): AK101 90mg on Week 0 and 4 administered subcutaneously followed by AK101 90mg administered subcutaneously every 12 weeks
  Interventions: Biological: AK101
- AK101 135mg -every 8 weeks (Experimental): AK101 135mg on Week 0 and 4 administered subcutaneously followed by AK101 135mg administered subcutaneously every 8 weeks
  Interventions: Biological: AK101
- AK101 135mg -every 12 weeks (Experimental): AK101 135mg on Week 0 and 4 administered subcutaneously followed by AK101 135mg administered subcutaneously every 12 weeks
  Interventions: Biological: AK101
- Placebo to AK101 (Placebo Comparator): Placebo on Week 0 and 4 administered subcutaneously followed by AK101 135mg administered subcutaneously at Week 12, 16 and then every 12 weeks
  Interventions: Biological: AK101; Biological: Placebo

INTERVENTIONS:
Biological: AK101 — an anti-IL-12/23p40 monoclonal antibody
Biological: Placebo — matching placebo
  Arms: Placebo to AK101

SUMMARY:
This is a multiple-center, randomized, double-blind, placebo-controlled Phase IIb study to evaluate the efficacy and safety of AK101, an anti-IL-12/23 p40 antibody, when administered subcutaneously, in subjects with moderate-to-severe plaque psoriasis. The study will consist of 3 periods: up to 4 weeks screening, 12 weeks double-blinded treatment and long-term follow-up period(up to 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Have had Plaque Psoriasis diagnosed at least 6 months prior to screening.
2. Clinical diagnosis of stable plaque psoriasis with involvement of ≥ 10% body surface area. Psoriasis area and severity index(PASI) ≥12. Physicians Global Assessment score ≥3.
3. Candidate for systemic therapy, defined as having psoriasis inadequately controlled by topical treatment (including topical corticosteroids) and/or phototherapy and/or previous systemic therapy.
4. Women of childbearing potential should not be in pregnancy or lactation, men and women of childbearing potential must agree to use adequate birth control measures during study participation and for 6 months after the last doses of study treatment.
5. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.

Exclusion Criteria:

1. Had nonplaque forms of psoriasis (e.g., Guttate, erythrodermic, or pustular).
2. Had other active skin diseases or skin infections (e.g., Bacterial, fungal or viral infection) that could affect psoriasis evaluation.
3. Had imaging diagnosis of pulmonary infection or fibrosis during the 3 months prior to screening.
4. History or evidence of active or latent tuberculosis at screening.
5. Serious systemic infections or local infections during the 2 months prior to screening.
6. History of cancer, including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin that have been excised and resolved).
7. Known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.
8. Known history of alcohol or drug abuse.
9. History or known presence of recurrent or chronic infection (e.g., hepatitis or C, human immunodeficiency virus [HIV], syphilis, TB).
10. Had received any DMARDs (e.g., Anti-malaria drug, retinoids, interferon, lithium) during 2 weeks prior to screening.
11. Had received any physical therapy (e.g., PUVA, ultra-violet therapy, tanning beds) during 2 weeks prior to screening.
12. Had received any systemic psoriasis therapy (e.g., Glucocorticoid, retinoids, ciclosporin, methotrexate, or tripterygium) during 4 weeks prior to screening.
13. Had enrolled in any other trials during 3 months prior to screening or concurrently enrolled in any other trials.
14. Had received previous treatment with any anti-IL-12/IL-23, IL-12, IL-23, IL-17 therapy for the treatment of psoriasis or psoriatic arthritis.
15. Had received natalizumab or any other drugs that regulate B cells or T cells (rituximab, abatacept, alemtuzumab) during 12 months prior to screening.
16. Had received other biologic therapy (e.g., TNF inhibitor) during 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieved ≥ 75% reduction in Psoriasis Area and Severity Index (PASI75) at Week 12 | Week 12
Incidence of treatment emergent adverse events (TEAEs) | From the time of signing the informed consent form till last follow-up visit (Up to Week 52)

SECONDARY OUTCOMES:
Number of participants who achieved ≥ 90% reduction in Psoriasis Area and Severity Index (PASI90) at Week 12 | At baseline and Week 12
Number of participants who achieved ≥ 75% reduction in Psoriasis Area and Severity Index (PASI75) | Up to Week 52 (except for Week 12)
Number of participants who achieved ≥ 90% reduction in Psoriasis Area and Severity Index (PASI90) | Up to Week 52( except for Week 12)
Number of participants who achieved 100% reduction in Psoriasis Area and Severity Index (PASI100) at Week 12 | Up to Week 52
Proportion of subjects who achieve a ≥ 4-point reduction in DLQI from baseline | Up to Week 52
  The DLQI is a dermatology-specific quality of life (QoL) instrument designed to assess the impact of the disease on a participant's QoL. It is a 10-item questionnaire that, in addition to evaluating overall Qol, can be used to assess six different aspects that mey affect QoL: 1) symptoms and feelings, 2) daily activities, 3) leisure, 4) work or school performance, 5) personal relationships, and 6) treatment.
Proportion of subjects who achieve Physician Global Assessment (PGA) of clear or almost clear (0 or 1) after treatment | Up to Week 52
Number of subjects who develop detectable anti-drug antibodies (ADAs) | Up to Week 52
  The immunogenicity of AK101 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)
Minimum observed concentration (Cmin) of AK101 at steady state | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, MD, Principal Investigator — Peking University People's Hospital; Hongzhong Jin, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No